CLINICAL TRIAL: NCT00001042
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Clinical Trial to Compare the Safety and Immunogenicity of Recombinant Envelope Protein rgp120/HIV-1SF2 (BIOCINE) Combined With Seven Adjuvants in Healthy HIV-1 Uninfected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 015; 10563 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Drug Therapy, Combination; Adjuvants, Immunologic; HIV Envelope Protein gp120; Acetylmuramyl-Alanyl-Isoglutamine; monophosphoryl lipid A; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Aluminum Hydroxide; monophosphoryl lipid A; Lipid A; Syntex adjuvant formulation; MF59 oil emulsion

INTERVENTIONS:
Biological: Aluminum hydroxide
Biological: Lipid A, Monophosphoryl
Biological: Lipid A, Liposome-encapsulated monophosphoryl
Biological: Syntex adjuvant formulation
Biological: MF59
Biological: Threonyl Muramyl Dipeptide
Biological: rgp120/HIV-1 SF-2
Biological: MTP-PE/MF59

SUMMARY:
To determine in healthy HIV-negative volunteers the safety and immunogenicity of rgp120/HIV-1SF2 (BIOCINE) formulated with each of seven adjuvants.

PER AMENDMENT 3/6/96: Purpose of the extension study - To determine the ability of immunization with rgp 120/SF-2 to induce an HIV-1 envelope-specific delayed-type hypersensitivity (DTH) response in volunteers who receive rsgp 120/MN skin testing.

One approach to improve the immunogenicity of an HIV-1 subunit protein vaccine is to combine the immunogen with an adjuvant. Adjuvants may augment vaccine immunogenicity by several mechanisms, and as a result induce a more favorable antibody response with high titers, which appear earlier in the course of immunization and persist over time.

DETAILED DESCRIPTION:
One approach to improve the immunogenicity of an HIV-1 subunit protein vaccine is to combine the immunogen with an adjuvant. Adjuvants may augment vaccine immunogenicity by several mechanisms, and as a result induce a more favorable antibody response with high titers, which appear earlier in the course of immunization and persist over time.

Volunteers are randomized to receive 50 mcg rgp120/HIV-1SF2 in combination with one of seven different adjuvants: aluminum hydroxide (alum), monophosphoryl lipid A, liposome-encapsulated monophosphoryl lipid A, MF59, MTP-PE/MF59, Syntex adjuvant formulation (SAF/2), and SAF/2 plus threonyl muramyl dipeptide (threonyl MDP). An additional placebo control arm of volunteers receive alum only. Doses are administered at 0, 2, and 6 months. Volunteers are followed for 1 year after the last immunization. Per 8/5/94 amendment, eligible volunteers except those who received monophosphoryl lipid A for the first three immunizations may receive a fourth dose at month 15.

PER AMENDMENT 3/6/96: Extension Study- Protocol 015 has been modified to add a special DTH study. At the end of the study, on day 784, intradermal injections of MN rsgp 120 will be administered to consenting volunteers who have received 4 immunizations as part of protocol 015. Follow up will be extended to 56 days after administration of the intradermal injections.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* HIV negativity by ELISA.
* Normal history and physical exam.
* CD4 count >= 400 cells/mm3.
* Lower risk sexual behavior.
* Normal urine dipstick with esterase and nitrite.

PER AMENDMENT 3/6/96:

* Extension study -
* Consenting Protocol 015 volunteers who have received four immunizations.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Hepatitis B surface antigen.
* Active syphilis. NOTE:Subjects for whom serology is documented to be a false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE:Subjects with a positive PPD and normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.
* Medical or psychiatric condition or occupational responsibilities that would preclude compliance.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, or autoimmune disease.
* History of anaphylaxis or other serious adverse reactions to vaccines.

PER AMENDMENT 3/6/96: Extension study -

* History of eczema or allergic-type reactions to vaccine in Protocol 015.

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days prior to study entry. (NOTE: Medically indicated subunit or killed vaccines, such as influenza or pneumococcal, are allowed but should be given at least 2 weeks prior to HIV immunizations.)
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.

PER AMENDMENT 3/6/96: Extension study -

* Use of systemic steroids in the past month.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within 6 months prior to study entry. Higher risk behavior for HIV infection (as determined by screening questionnaire), including history of injection drug use within the last 12 months and higher or intermediate risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Study Completion 1996-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: McElrath J, Study Chair
Locations (3):
- United States (3):
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Zolla-Pazner S, Alving C, Belshe R, Berman P, Burda S, Chigurupati P, Clements ML, Duliege AM, Excler JL, Hioe C, Kahn J, McElrath MJ, Sharpe S, Sinangil F, Steimer K, Walker MC, Wassef N, Xu S. Neutralization of a clade B primary isolate by sera from human immunodeficiency virus-uninfected recipients of candidate AIDS vaccines. J Infect Dis. 1997 Apr;175(4):764-74. doi: 10.1086/513969. PMID 9086128